CLINICAL TRIAL: NCT01962103
Title: A Phase 1/2, Multicenter, Open-label, Dose-finding Study to Assess the Safety, Tolerability, and Preliminary Efficacy of Weekly Nab-paclitaxel in Pediatric Patients With Recurrent or Refractory Solid Tumors.
Brief Title: Study to Find a Safe Dose and Show Early Clinical Activity of Weekly Nab-paclitaxel in Pediatric Patients With Recurrent/ Refractory Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABI-007-PST-001
Record Dates: First submitted 2013-09-27; First posted 2013-10-14 (Estimated); Results first posted 2018-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Neuroblastoma; Rhabdomyosarcoma; Ewing's Sarcoma; Ewing's Tumor; Sarcoma, Ewing's; Sarcomas, Epitheliod; Sarcoma, Soft Tissue; Sarcoma, Spindle Cell; Melanoma; Malignant Melanoma; Clinical Oncology; Oncology, Medical; Pediatrics, Osteosarcoma; Osteogenic Sarcoma; Osteosarcoma Tumor; Sarcoma, Osteogenic; Tumors; Cancer; Neoplasia; Neoplasm; Histiocytoma; Fibrosarcoma; Dermatofibrosarcoma
Keywords: Neuroblastoma; Rhabdomyosarcoma; Soft Tissue; Pediatric Oncology; Abraxane; albumin-bound paclitaxel; nab-paclitaxel; ABI-007; taxane; solid tumors
MeSH Terms: conditions — Neuroblastoma; Rhabdomyosarcoma; Sarcoma, Ewing; Sarcoma; Melanoma; Neoplasms; Osteosarcoma; Histiocytoma; Fibrosarcoma; Dermatofibrosarcoma | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- nab-paclitaxel (Experimental): nab-paclitaxel 100-240 mg/m2 IV on Days 1, 8 and 15 of a 28-day cycle.
  Interventions: Drug: nab-paclitaxel
- Phase 1: Nab-Paclitaxel 120 mg/m^2 (Experimental): nab-paclitaxel 120 mg/m^2 IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity to establish the RP2D.
  Interventions: Drug: nab-paclitaxel
- Phase 1: Nab-Paclitaxel 150 mg/m^2 (Experimental): nab-paclitaxel 150 mg/m^2 IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity to establish the RP2D.
  Interventions: Drug: nab-paclitaxel
- Phase 1: Nab-Paclitaxel 180 mg/m^2 (Experimental): nab-paclitaxel 180 mg/m^2 IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity to establish the RP2D.
  Interventions: Drug: nab-paclitaxel
- Phase 1: Nab-Paclitaxel 210 mg/m^2 (Experimental): nab-paclitaxel 210 mg/m^2 IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity to establish the RP2D.
  Interventions: Drug: nab-paclitaxel
- Phase 1: Nab-Paclitaxel 240 mg/m^2 (Experimental): nab-paclitaxel 240 mg/m^2 IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity to establish the RP2D.
  Interventions: Drug: nab-paclitaxel
- Phase 1: Nab-Paclitaxel 270 mg/m^2 (Experimental): nab-paclitaxel 270 mg/m^2 IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity to establish the RP2D.
  Interventions: Drug: nab-paclitaxel
- Phase 2: Ewing's Sarcoma (Experimental): Participants with Ewing's sarcoma: nab-paclitaxel at the RP2D (240 mg/m^2 in participants weighing > 10 kg and 11.5 mg/kg in participants weighing ≤ 10 kg) IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity.
  Interventions: Drug: nab-paclitaxel
- Phase 2: Neuroblastoma (Experimental): Participants with neuroblastoma: nab-paclitaxel at the RP2D (240 mg/m^2 in participants weighing > 10 kg and 11.5 mg/kg in participants weighing ≤ 10 kg) IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity.
  Interventions: Drug: nab-paclitaxel
- Phase 2: Rhabdomyosarcoma (Experimental): Participants with rhabdomyosarcoma: nab-paclitaxel at the RP2D (240 mg/m^2 in participants weighing > 10 kg and 11.5 mg/kg in participants weighing ≤ 10 kg) IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity.
  Interventions: Drug: nab-paclitaxel

INTERVENTIONS:
Drug: nab-paclitaxel — nab-paclitaxel 120-270 mg/m2 IV on Days 1, 8 and 15 of a 28-day cycle
  Other Names: Abraxane
  Arms: nab-paclitaxel
Drug: nab-paclitaxel — IV infusion
  Other Names: Abraxane
  Arms: Phase 1: Nab-Paclitaxel 120 mg/m^2; Phase 1: Nab-Paclitaxel 150 mg/m^2; Phase 1: Nab-Paclitaxel 180 mg/m^2; Phase 1: Nab-Paclitaxel 210 mg/m^2; Phase 1: Nab-Paclitaxel 240 mg/m^2; Phase 1: Nab-Paclitaxel 270 mg/m^2; Phase 2: Ewing's Sarcoma; Phase 2: Neuroblastoma; Phase 2: Rhabdomyosarcoma

SUMMARY:
The purpose of this study is to find the safe dose of nab-paclitaxel in children with solid tumors, and to see if it works to treat these solid tumors in children and young adults (in Phase 1 ≤ 18 years old and in Phase 2 ≤ 24 years old). After the final dose has been chosen, patients will be enrolled according to the specific solid tumor type, (neuroblastoma, rhabdomyosarcoma, or Ewing's sarcoma), to see how nab-paclitaxel works in treating these tumors.

DETAILED DESCRIPTION:
ABI-007-PST-001 is a Phase 1/2, multicenter, open-label, dose-finding study to assess the safety , tolerability, and preliminary efficacy of weekly nab-paclitaxel in pediatric patients with recurrent or refractory solid tumors (excluding brain tumors). The Phase 1 portion of the study, with a dose escalation design, ended and the recommended Phase 2 dose (RP2D) was determined as 240 mg/m^2 intravenously (IV) in patients weighing > 10 kg and 11.5 mg/kg in patients weighing ≤ 10 kg, on Days 1, 8 and 15 of a 28-day cycle. The Phase 2 portion of the study will enroll additional patients at the RP2D into 1 of 3 solid tumor groups [neuroblastomas, rhabdomyosarcomas, Ewing's sarcomas]. Both phases of the study are open-label and conducted at multiple centers.

The Phase 2 is using a Simon 2-stage design to monitor patient enrollment for each group separately. The rhabdomyosarcoma group, neuroblastoma or Ewing's sarcoma groups did not reach the expected number of 2 responders out of 14 efficacy eligible patients. Consequently, the groups were stopped.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be enrolled in the study:

  1. Patient has a confirmed solid tumor diagnosis according to the

     following:
     1. Phase 1: patient has a recurrent or refractory solid tumor that has

        progressed or did not respond to standard therapy, or for which no

        standard anticancer therapy exists
     2. Phase 2: patient has radiologically documented measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 (for neuroblastoma, evaluable disease by 123^I-metaiodobenzylguanidine [MIBG]/Curie score is also acceptable) in 1 of the following tumor types and has failed up to 3 lines of treatment: Group 1: neuroblastoma, Group 2: rhabdomyosarcoma; Group 3: Ewing's sarcoma.
  2. The patient has a Lansky/Karnofsky performance status score of ≥ 70%.
  3. The patient has adequate serum chemistry levels, evidenced by the

     following laboratory values
     1. aspartate aminotransferase (AST)/serum glutamic-oxaloacetric

        transaminase (SGOT), alanine aminotransferase (ALT)/serum glutamic

        pyruvate transaminase (SGPT) ≤ 2.5 × upper limit of normal range (ULN)
     2. Total bilirubin ≤ 1.5 × ULN
     3. Creatinine ≤ 1.5 × ULN
  4. The patient has adequate bone marrow function, evidenced by the

     following:
     1. Absolute neutrophil count ≥ 1.0 × 10^9 cells/L
     2. Platelets ≥ 80 × 10^9 cells/L (transfusion independent, defined as not

        receiving platelet transfusions within 7 days prior to laboratory sample). In the phase 2 portion, for patients with known bone marrow involvement, platelets ≥ 50 × 10^9 cells/L
     3. Hemoglobin ≥ 8 g/dL (transfusion is permitted to fulfill this criterion).
  5. The patient (when applicable) or patient's parent(s) or legal guardian(s)

     understand(s) and voluntarily signed an informed consent document prior

     to any study-related assessments/procedures being conducted. Where

     locally applicable, the patient also understands and voluntarily provides

     his/her assent prior to any study-related assessments/procedures being

     conducted.
  6. Male patients of childbearing potential must use a condom during

     sexual intercourse and shall not father a child during the study and for 6 months after the last dose of study medication.
  7. Female patients of childbearing potential [defined as all female

     patients ≥ 12 years old or who have reached menarche, whichever occurs

     first] must have both of the following:

     a. Agree to the use of two physician-approved contraceptive methods

     simultaneously or practice complete abstinence while on study medication or for a longer period if required by regulations.

     i. True abstinence: When this is in line with the preferred and usual

     lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation,

     symptothermal, postovulation methods) and withdrawal are not

     acceptable methods of contraception.

     ii. Acceptable contraceptive methods include: oral, injectable, or

     implantable hormonal contraceptive; tubal ligation; intra-uterine device;

     barrier contraceptive with spermicide; or vasectomized partner) including

     at least one barrier method.

     b. Have negative serum pregnancy test result at screening confirmed by

     negative urine pregnancy dipstick within 72 hours prior to first dose of

     investigational product (if serum test occurred > 72 hours from first

     dose); pregnancy test with sensitivity of at least 25 mIU/mL.

     Exclusion Criteria:
     * The presence of any of the following will exclude a patient from enrollment:

  <!-- -->

  1. The patient has a primary brain tumor(s) or brain metastasis (unless metastasis is treated and stable for > 28 days). In patients who are symptomatic, a brain scan is required to exclude metastasis.
  2. The patient has received therapeutic dose chemotherapy or radiotherapy ≤ 21 days prior to start of investigational product.
  3. The patient has received maintenance dose chemotherapy (e.g., low dose cyclophosphamide) ≤ 7 days from the first dose of investigational product.
  4. The patient has received any investigational therapy ≤ 28 days prior to start of investigational product. Investigational therapy is defined as any medicinal product that is not approved in the country of treatment for any indication, adult or pediatric.
  5. The patient has received any biological therapy ≤ 7 days prior to the start of investigational product, or monoclonal antibody ≤ 3 half-lives or 28 days, whichever is shorter, prior to the first dose of investigational product.
  6. The patient has received any hematopoietic stem cell transplantation (HSCT) ≤ 3 months prior to start of investigational product.
  7. The patient has received allogeneic hematopoietic stem cell transplantation (HSCT) ≤ 3 months or autologous HSCT ≤ 21 days prior to start of investigational product.
  8. The patient has not recovered from the acute toxic effects of prior chemotherapy, radiation, or major surgery/significant trauma.
  9. The patient has had minor surgery ≤ 7 days from the start of study treatment (excluding the placement of central/peripheral lines, skin biopsy).
  10. The patient has a known history of stroke, myocardial infarction, peripheral vascular disease, or recent (within 3 months) uncontrolled deep venous thrombosis.
  11. The patient has a known history or current diagnosis of human immunodeficiency virus (HIV) infection, regardless of treatment status.
  12. The patient has an uncontrolled intercurrent illness including but not limited to ongoing or active infection requiring antibiotic, antifungal, or antiviral therapy, symptomatic heart failure, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
  13. The patient has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from participating in the study.
  14. The patient has any condition, including the presence of laboratory abnormalities, that places the patient at unacceptable risk if he/she were to participate in the study.
  15. The patient has any condition that confounds the ability to interpret data from the study.
  16. The patient or parent(s)/guardian(s) is/are unable to comply with the study visit schedule and other protocol requirements, in the opinion of the investigator.
  17. The patient has ≥ Grade 2 peripheral neuropathy by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) at screening.

Ages: 6 Months to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 107 (Actual)
Dates: Start 2013-12-04 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ileana Elias, M.D., Study Director — Celgene Corporation
Locations (20):
- United States (2):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Columbia University Medical Center, New York, New York
- The Hospital for Sick Children, Toronto, Ontario, Canada
- France (4):
  - Institute for Pediatric Hematology - Oncology, Leon Berard Cancer Center, Lyon
  - Hopital d'Enfants, CHU Nancy, Nancy
  - Institut Curie, Paris
  - Institut Gustave Roussy, Villejuif
- Italy (6):
  - Azienda Ospedaliera Universitaria Meyer, Florence
  - Children's Hospital Largo, Genova
  - Istituto Nazionale Tumori, Milan
  - Clinica di Oncoematologia, Padua
  - Policlinico Agostino Gemelli, Rome
  - l'Azienda Ospedaliera Regina Margherita - Sant Anna, Torino
- Spain (5):
  - Hospital Universitario Vall D Hebron, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
  - Spanish National Cancer Research Centre, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Unidad de Oncologia Pediatrica, Hospital Universitario la Fe, Valencia
- Universitäts-Kinderklinik, Zurich, Switzerland
- Royal Marsden Hospital, Sutton, United Kingdom

REFERENCES:
- [Background] Moreno L, Casanova M, Chisholm JC, Berlanga P, Chastagner PB, Baruchel S, Amoroso L, Gallego Melcon S, Gerber NU, Bisogno G, Fagioli F, Geoerger B, Glade Bender JL, Aerts I, Bergeron C, Hingorani P, Elias I, Simcock M, Ferrara S, Le Bruchec Y, Slepetis R, Chen N, Vassal G. Phase I results of a phase I/II study of weekly nab-paclitaxel in paediatric patients with recurrent/refractory solid tumours: A collaboration with innovative therapies for children with cancer. Eur J Cancer. 2018 Sep;100:27-34. doi: 10.1016/j.ejca.2018.05.002. Epub 2018 Jun 21. PMID 29936064
- [Derived] Amoroso L, Castel V, Bisogno G, Casanova M, Marquez-Vega C, Chisholm JC, Doz F, Moreno L, Ruggiero A, Gerber NU, Fagioli F, Hingorani P, Melcon SG, Slepetis R, Chen N, le Bruchec Y, Simcock M, Vassal G. Phase II results from a phase I/II study to assess the safety and efficacy of weekly nab-paclitaxel in paediatric patients with recurrent or refractory solid tumours: A collaboration with the European Innovative Therapies for Children with Cancer Network. Eur J Cancer. 2020 Aug;135:89-97. doi: 10.1016/j.ejca.2020.04.031. Epub 2020 Jun 15. PMID 32554315
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixty-five participants were included in the Phase 1 enrolled population, and 64 enrolled partcipants received at least 1 dose of study drug and were included in the safety population, noted below. Forty-two participants were included in the Phase 2 enrolled and safety populations.
Groups:
- Phase 1: Nab-Paclitaxel 120 mg/m^2: nab-paclitaxel 120 mg/m^2 intravenously (IV) on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity to establish the recommended phase 2 dose (RP2D).
Period: Phase 1
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2 | Phase 2: Ewing's Sarcoma | Phase 2: Neuroblastoma | Phase 2: Rhabdomyosarcoma
Started | 16 | 8 | 14 | 11 | 8 | 7 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 8 | 14 | 11 | 8 | 7 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 2 | 1 | 2 | 2 | 0 | 0 | 0
Not completed — Progressive Disease | 8 | 6 | 8 | 4 | 5 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Symptomatic Deterioration | 3 | 2 | 2 | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Miscellaneous | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2 | Phase 2: Ewing's Sarcoma | Phase 2: Neuroblastoma | Phase 2: Rhabdomyosarcoma
Started | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 14 | 14
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 (completed treatment) | 0 (completed treatment) | 0 (completed treatment)
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 14 | 14
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 12 | 11
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2 | Phase 2: Ewing's Sarcoma | Phase 2: Neuroblastoma | Phase 2: Rhabdomyosarcoma | Total
Number analyzed (Participants) | 16 | 8 | 14 | 11 | 8 | 7 | 14 | 14 | 14 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (3.32) | 12.1 (5.84) | 10.2 (4.64) | 10.2 (5.36) | 11.6 (4.63) | 12.1 (2.97) | 10.1 (4.63) | 7.1 (3.42) | 12.4 (6.42) | 10.7 (4.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 9 | 7 | 1 | 3 | 6 | 5 | 9 | 53
  Male | 7 | 4 | 5 | 4 | 7 | 4 | 8 | 9 | 5 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 1 | 1 | 3 | 0 | 0 | 2 | 5 | 17
  Not Hispanic or Latino | 6 | 5 | 7 | 10 | 5 | 5 | 11 | 8 | 8 | 65
  Unknown or Not Reported | 8 | 0 | 6 | 0 | 0 | 2 | 3 | 4 | 1 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 8 | 9 | 9 | 8 | 5 | 11 | 11 | 12 | 84
  Not Collected or Reported | 5 | 0 | 5 | 0 | 0 | 1 | 3 | 3 | 1 | 18
  Other, Not Specified | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 3
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Participants With Any Prior Cancer Treatment [Count of Participants; unit: Participants]
  Any Prior Cancer Treatment | 16 | 8 | 14 | 11 | 8 | 7 | 14 | 14 | 14 | 106
  Prior Radiation Therapy | 9 | 4 | 11 | 7 | 6 | 6 | 12 | 10 | 10 | 75
  Prior Cancer Surgeries | 14 | 7 | 9 | 9 | 5 | 7 | 10 | 11 | 6 | 78
  Prior Systemic Anticancer Therapy | 16 | 8 | 14 | 11 | 8 | 7 | 14 | 14 | 14 | 106
  Prior Systemic Anticancer Regimens | 16 | 8 | 14 | 11 | 8 | 7 | 14 | 14 | 14 | 106
  Prior Stem Cell Transplants | 2 | 2 | 3 | 2 | 3 | 2 | 3 | 10 | 0 | 27
  Other Prior Anticancer Therapies | 2 | 0 | 1 | 3 | 2 | 0 | 1 | 6 | 0 | 15
Number of Prior Systemic Anticancer Regimens Received [Mean (Standard Deviation); unit: systemic anticancer regimens] | 3.69 (1.815) | 3.25 (1.832) | 3.64 (1.946) | 3.64 (2.461) | 3.00 (1.309) | 3.00 (0.816) | 2.50 (0.519) | 2.14 (0.663) | 2.21 (0.579) | 2.99 (1.552)

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as investigational product (IP)-related adverse events occurring during the DLT assessment period that led to treatment discontinuation or met one of the following criteria: - Common Terminology Criteria for Adverse Events (CTCAE) Grade (Gr) 3 or 4 nonhematologic toxicity (excluding transient transaminitis) - CTCAE Gr 3 or 4 nausea or vomiting that persisted > 5 days despite maximal anti-emetic treatment - CTCAE Gr 4 thrombocytopenia or anemia that persisted > 7 days or required transfusion > 7 days - CTCAE Gr 3 thrombocytopenia with bleeding - CTCAE Gr 4 uncomplicated neutropenia lasting > 7 days - Febrile neutropenia with confirmed bacterial infection - CTCAE Gr 3 hematologic toxicity requiring treatment (tx) delay > 21 days. Use of "..." in the table rows signifies the continuation of row title per the above list.
Time Frame: DLT assessment period: For participants > 10 kg: the first 28-day cycle including Cycle 2 Day 1 predose evaluations; for participants ≤ 10 kg: the first two 28-day cycles including Cycle 3 Day 1 predose evaluations
Population: Dose Determining Set (DDS): all Phase 1 participants who received all 3 weekly doses of nab-paclitaxel at the cohort planned dose during Cycle 1 and had adequate safety assessments during the DLT assessment period or experienced a DLT. The DDS did not include participants who were enrolled at each dose once the dose had been determined to be safe.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 7
Participants
  At least 1 DLT | 1 | 0 | 0 | 0 | 0 | 1
  Gr 3/4 Nonhematologic Toxicity... | 1 | 0 | 0 | 0 | 0 | 0
  Gr 3/4 Nausea or Vomiting Persisting >5 days... | 0 | 0 | 0 | 0 | 0 | 0
  Gr 4 Thrombocytopenia/Anemia Persisting >7 days... | 0 | 0 | 0 | 0 | 0 | 0
  Gr 3 Thrombocytopenia with Bleeding | 0 | 0 | 0 | 0 | 0 | 0
  Gr 4 Uncomplicated Neutropenia Lasting >7 days | 0 | 0 | 0 | 0 | 0 | 1
  Febrile Neutropenia+Confirmed Bacterial Infection | 0 | 0 | 0 | 0 | 0 | 0
  Gr3 Hematologic Toxicity Requiring Tx Delay... | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Phase 1: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. A serious AE (SAE) is any AE occurring at any dose that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. TEAEs were defined as AEs that began or worsened in severity on or after the date of the first dose of study drug and within 28 days of the date of the last dose of study drug. The severity of an AE was graded according to the CTCAE, Version 4.0.
Time Frame: Median treatment duration in Phase 1 was 7.0 weeks, with minimum and maximum duration of 1 and 49 weeks, respectively. Participants were followed for 28 days after discontinuing treatment for safety and monitoring of AEs.
Population: Safety Population: all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 16 | 8 | 14 | 11 | 8 | 7
Participants
  TEAE | 16 | 8 | 14 | 11 | 8 | 7
  Treatment-related (TR) TEAE | 14 | 8 | 12 | 11 | 7 | 7
  Grade 3 or 4 TEAE | 13 | 8 | 10 | 10 | 8 | 7
  TR Grade 3 or 4 TEAE | 9 | 7 | 7 | 9 | 7 | 7
  Serious TEAE | 10 | 7 | 6 | 5 | 3 | 4
  TR Serious TEAE | 1 | 4 | 4 | 2 | 1 | 3
  TEAE Leading to Drug Discontinuation | 4 | 0 | 2 | 1 | 2 | 2
  TR TEAE Leading to Drug Discontinuation | 1 | 0 | 0 | 1 | 2 | 2
  TEAE Leading to Dose Reduction | 0 | 1 | 2 | 1 | 3 | 3
  TR TEAE Leading to Dose Reduction | 0 | 1 | 2 | 1 | 3 | 3
  TEAE Leading to Drug Interruption | 2 | 2 | 3 | 4 | 3 | 2
  TR TEAE Leading to Drug Interruption | 0 | 2 | 1 | 3 | 3 | 2
  TEAE Leading to Death | 2 | 1 | 0 | 0 | 1 | 1
  TR TEAE Leading to Death | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase 2: Overall Response Rate (ORR)
Description: Overall response rate was defined as the percentage of participants who achieved a complete response (CR; disappearance of all target lesions) or partial response (PR; at least a 30% decrease in the sum of diameters of target lesions) confirmed no less than 4 weeks after the criteria for response were first met using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 guidelines. (For Phase 2 neuroblastoma participants who had both RECIST and Curie Score tumor evaluations, both tumor response results were considered and an overall response was derived.) Confidence interval was obtained using the Clopper-Pearson method.
Time Frame: Median treatment duration in Phase 2 per group: Ewings Sarcoma = 14 weeks (3-31), Neuroblastoma = 7 weeks (3-23), Rhabdomyosarcoma = 5 weeks (1-13).
Population: Efficacy Evaluable Population: participants who met eligibility criteria for Phase 2, completed at least 1 dose of study drug, and had baseline and at least 1 postbaseline efficacy assessment if having not discontinued the investigational product prior to postbaseline efficacy assessment due to disease progression or systematic deterioration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ewing's Sarcoma | Phase 2: Neuroblastoma | Phase 2: Rhabdomyosarcoma
Number analyzed (Participants) | 13 | 14 | 14
percentage of participants | 0 [0.0 to 24.7] | 0 [0.0 to 23.2] | 7.1 [0.2 to 33.9]

4. Secondary Outcome: Phase 1: ORR
Description: Overall response rate was defined as the percentage of participants who achieved a complete response (CR; disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions) confirmed no less than 4 weeks after the criteria for response were first met) using RECIST version 1.1 guidelines over the total number of participants available for the analysis. Confidence interval was obtained using the Clopper-Pearson method.
Time Frame: Median treatment duration in Phase 1 was 7.0 weeks, with minimum and maximum duration of 1 and 49 weeks, respectively.
Population: Efficacy Evaluable Population: participants who met eligibility criteria for Phase 1, completed at least 1 dose of study drug, and had baseline and at least 1 postbaseline efficacy assessment if having not discontinued the investigational product prior to postbaseline efficacy assessment due to disease progression or systematic deterioration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 14 | 8 | 12 | 10 | 8 | 7
percentage of participants | 0 [0.0 to 23.2] | 0 [0.0 to 36.9] | 0 [0.0 to 26.5] | 0 [0.0 to 30.8] | 12.5 [0.3 to 52.7] | 14.3 [0.4 to 57.9]

5. Secondary Outcome: Phase 1: Maximum Observed Concentration of Paclitaxel in Blood Plasma (Cmax)
Time Frame: Cycle 1 Day 1 (Participants ≥ 6 years: 1-2 minutes prior to the end of infusion [EOI], and 15 minutes, 1, 3, 5, 8, 24, 48, and 72 hours after the EOI. Participants <6 years: 1-2 minutes prior to the EOI, and 15 minutes, 3, 5, and 24 hours after the EOI.)
Population: Pharmacokinetic (PK) population: all participannts who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 13 | 7 | 12 | 9 | 7 | 6
ng/mL | 3488 (73.7) | 5468 (38.0) | 5597 (33.4) | 5616 (63.9) | 7831 (23.1) | 8078 (41.5)

6. Secondary Outcome: Phase 1: Cmax - Dose-Normalized
Time Frame: as for outcome 5
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/[mg]
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 13 | 7 | 12 | 9 | 7 | 6
ng/mL/[mg] | 23.3 (87.5) | 25.4 (46.6) | 27.3 (47.3) | 23.2 (80.3) | 28.2 (48.7) | 21.0 (46.6)

7. Secondary Outcome: Phase 1: Area Under the Plasma Concentration-Time Curve (AUC)
Description: Measurements include: AUC from time zero to the last measurable concentration (AUCt), AUC from time zero to 24 hours (AUC24), and AUC from time zero to infinity (AUCinf).
Time Frame: as for outcome 5
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data for given measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 13 | 7 | 12 | 9 | 7 | 6
ng*h/mL
  AUCt | 7844 (73.4) | 10374 (91.8) | 9690 (37.1) | 11817 (64.0) | 12706 (29.2) | 11245 (22.6)
  AUC24: number analyzed (Participants) | 13 | 7 | 12 | 8 | 7 | 6
  AUC24 | 6392 (79.0) | 8944 (85.9) | 8365 (37.7) | 10932 (66.3) | 11167 (27.4) | 9768 (20.7)
  AUCinf: number analyzed (Participants) | 9 | 6 | 10 | 6 | 6 | 5
  AUCinf | 8867 (85.4) | 11992 (99.8) | 10087 (38.4) | 14361 (72.1) | 14242 (29.2) | 12424 (28.5)

8. Secondary Outcome: Phase 1: AUC - Dose-Normalized
Description: Measurements include: AUC24 and AUCinf.
Time Frame: as for outcome 5
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/[mg]
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 13 | 7 | 12 | 8 | 7 | 6
ng*h/mL/[mg]
  AUC24 | 42.7 (77.4) | 41.6 (87.0) | 40.8 (39.7) | 43.3 (63.6) | 40.2 (65.4) | 25.4 (26.1)
  AUCinf: number analyzed (Participants) | 9 | 6 | 10 | 6 | 6 | 5
  AUCinf | 62.0 (75.7) | 49.2 (101) | 47.8 (39.8) | 64.8 (25.4) | 52.3 (67.4) | 31.3 (34.9)

9. Secondary Outcome: Phase 1: Clearance (CL)
Description: Measurement of renal clearance from the body.
Time Frame: as for outcome 5
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 9 | 6 | 10 | 6 | 6 | 5
L/h | 16.1 (75.6) | 20.3 (101) | 20.9 (39.9) | 15.4 (25.4) | 19.1 (67.4) | 31.9 (35.0)

10. Secondary Outcome: Phase 1: CL - Body Surface Area (BSA)-Normalized
Description: Measurement of renal clearance from the body.
Time Frame: as for outcome 5
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h/m^2
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 9 | 6 | 10 | 6 | 6 | 5
L/h/m^2 | 13.5 (85.1) | 12.5 (99.3) | 17.8 (38.3) | 14.6 (72.3) | 16.7 (29.2) | 21.8 (28.4)

11. Secondary Outcome: Phase 1: Volume of Distribution (Vss)
Time Frame: as for outcome 5
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 9 | 6 | 10 | 6 | 6 | 5
liters | 127 (145) | 266 (78.3) | 146 (106) | 89.8 (45.1) | 175 (117) | 446 (17.6)

12. Secondary Outcome: Phase 1: Vss - BSA-Normalized
Time Frame: as for outcome 5
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/m^2
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2
Number analyzed (Participants) | 9 | 6 | 10 | 6 | 6 | 5
L/m^2 | 106 (95.3) | 164 (78.4) | 124 (82.8) | 84.9 (49.7) | 154 (56.5) | 304 (29.0)

13. Secondary Outcome: Phase 1 and 2 Population PK: Volume of Distribution of the Central Compartment (V1)
Description: Population PK analysis was performed using nonlinear mixed effect modeling. The estimated allometric function for V1 was 0.888.
Time Frame: Cycle 1 Day 1 (Participants ≥ 6 years: 1-2 minutes prior to the end of infusion [EOI], and 15 minutes, 1, 3, 5, 8, 24, 48, and 72 hours after the EOI. Participants < 6 years: 1-2 minutes prior to the EOI, and 15 minutes, 3, 5, and 24 hours after the EOI.)
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Number; unit: liters
Groups:
- PK Population: Phase 1: nab-paclitaxel 120-270 mg/m^2 IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity to establish the RP2D. Phase 2: nab-paclitaxel at the RP2D (240 mg/m^2 in participants weighing > 10 kg and 11.5 mg/kg in participants weighing ≤ 10 kg) IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity.
Arm/Group | PK Population
Number analyzed (Participants) | 106
liters | 11.8

14. Secondary Outcome: Phase 1 and 2 Population PK: Maximum Elimination Rate From the Central Compartment (VMEL)
Description: Population PK analysis was performed using nonlinear mixed effect modeling. The estimated allometric function for VMEL was 1.12.
Time Frame: as for outcome 13
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data
Measure: Number; unit: μg/h
Groups:
- PK Population: The PK population included all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Arm/Group | PK Population
Number analyzed (Participants) | 106
μg/h | 31983

15. Secondary Outcome: Phase 1 and 2 Population PK: Concentration in the Central Compartment at 50% of VMEL (KMEL)
Description: Population PK analysis was performed using nonlinear mixed effect modeling.
Time Frame: as for outcome 13
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data
Measure: Number; unit: μg/L
Arm/Group | PK Population
Number analyzed (Participants) | 106
μg/L | 951

16. Secondary Outcome: Phase 1 and 2 Population PK: Intercompartmental CL Between the Central Compartment and the First Peripheral Compartment (Q2)
Description: Population PK analysis was performed using nonlinear mixed effect modeling. The estimated allometric function for Q2 was 1.12.
Time Frame: as for outcome 13
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Number; unit: L/h
Arm/Group | PK Population
Number analyzed (Participants) | 106
L/h | 22.4

17. Secondary Outcome: Phase 1 and 2 Population PK: Intercompartmental CL Between the Central Compartment and the Second Peripheral Compartment (Q3)
Description: Population PK analysis was performed using nonlinear mixed effect modeling. The estimated allometric function for Q3 was 1.12.
Time Frame: as for outcome 13
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Number; unit: L/h
Arm/Group | PK Population
Number analyzed (Participants) | 106
L/h | 34.8

18. Secondary Outcome: Phase 1 and 2 Population PK: Volume of Distribution of the First Peripheral Compartment (V2)
Description: Population PK analysis was performed using nonlinear mixed effect modeling. The estimated allometric function for V2 was 0.888.
Time Frame: as for outcome 13
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Number; unit: liters
Arm/Group | PK Population
Number analyzed (Participants) | 106
liters | 545

19. Secondary Outcome: Phase 1 and 2 Population PK: Volume of Distribution of the Second Peripheral Compartment (V3)
Description: Population PK analysis was performed using nonlinear mixed effect modeling. The estimated allometric function for V3 was 0.888.
Time Frame: as for outcome 13
Population: PK population: all participants who received at least one dose of nab-paclitaxel and had evaluable concentration data.
Measure: Number; unit: liters
Arm/Group | PK Population
Number analyzed (Participants) | 106
liters | 45.3

20. Secondary Outcome: Phase 2: Duration of Response (DOR)
Description: Duration of response was defined as the time from the date of the first response (CR/PR, using RECIST version 1.1 guidelines) to disease progression for participants with a confirmed CR or PR. Participants who did not have disease progression or had not died were censored at the time of their last disease assessment or at time of start of new anticancer therapy, whichever occurred first. (For Phase 2 neuroblastoma patients who had both RECIST version 1.1 and Curie Score tumor evaluations, both tumor responses results were considered and an overall response was derived.)
Time Frame: Median treatment duration in Phase 2 per group: Ewings Sarcoma = 14 weeks (3-31), Neuroblastoma = 7 weeks (3-23), Rhabdomyosarcoma = 5 weeks (1-13). Participants were followed until disease progression (if applicable) up to a maximum of 100.3 weeks.
Population: Efficacy Evaluable Population: participants (with response) who met eligibility criteria for Phase 2, completed ≥ 1 dose of study drug, and had baseline and ≥ 1 postbaseline efficacy assessment if having not discontinued the investigational product prior to postbaseline efficacy assessment due to disease progression or systematic deterioration.
Measure: Median (Full Range); unit: weeks
Arm/Group | Phase 2: Ewing's Sarcoma | Phase 2: Neuroblastoma | Phase 2: Rhabdomyosarcoma
Number analyzed (Participants) | 0 | 0 | 1
weeks |  |  | 6.14 [6.14 to 6.14]

21. Secondary Outcome: Phase 2: Disease Control Rate (DCR)
Description: Disease control rate was defined as the percentage of participants who achieved either a stable disease maintained for ≥ 16 weeks or confirmed CR (confirmed no less than 4 weeks after criteria for response were first met) or confirmed PR (confirmed no less than 4 weeks after criteria for response were first met) over the total number of participants available for the analysis. Confidence interval was obtained using the Clopper-Pearson method.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ewing's Sarcoma | Phase 2: Neuroblastoma | Phase 2: Rhabdomyosarcoma
Number analyzed (Participants) | 13 | 14 | 14
percentage of participants | 30.8 [9.1 to 61.4] | 7.1 [0.2 to 33.9] | 7.1 [0.2 to 33.9]

22. Secondary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the first dose date to the start of disease progression or participant death (any cause), whichever occurred first. Disease progression was classed as either a disease progression observed as a response assessment, or a disease progression or symptomatic deterioration at treatment/study discontinuation. Participants who did not have disease progression or had not died were censored at the last known time that the participant was progression free. Disease progression was considered according to RECIST version 1.1 for Phase 2 Ewing's sarcoma and rhabdomyosarcoma participants. (For Phase 2 neuroblastoma participants who had both RECIST 1.1 and Curie score tumor evaluations, both tumor responses results were considered and an overall response was derived.) Median PFS time was estimated through Kaplan-Meier methods. 95% confidence interval about the median time to PFS event was obtained using Greenwood's method.
Time Frame: as for outcome 20
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Ewing's Sarcoma | Phase 2: Neuroblastoma | Phase 2: Rhabdomyosarcoma
Number analyzed (Participants) | 13 | 14 | 14
weeks | 13 [7.4 to 16.1] | 7.4 [4.6 to 8.1] | 5.1 [2.1 to 7.9]

23. Secondary Outcome: Phase 2: Kaplan-Meier Estimate of Overall Survival Rate at 1 Year
Description: Overall survival was defined as the time from the first dose date to date of death (any cause). Participants who were alive were censored at the last known time that the participant was alive.
Time Frame: 1 year
Population: Efficacy Evaluable Population: participants who met eligibility criteria for Phase 2, completed ≥1 dose of study drug, and had baseline and ≥1 postbaseline efficacy assessment if having not discontinued the investigational product prior to postbaseline efficacy assessment due to disease progression or systematic deterioration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ewing's Sarcoma | Phase 2: Neuroblastoma | Phase 2: Rhabdomyosarcoma
Number analyzed (Participants) | 13 | 14 | 14
percentage of participants | 48 [14 to 76] | 25 [4 to 54] | 15 [2 to 39]

24. Secondary Outcome: Phase 2: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. A SAE is any AE occurring at any dose that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. TEAEs were defined as AEs that began or worsened in severity on or after the date of the first dose of study drug and within 28 days of the date of the last dose of study drug. The severity of the AEs was graded according to the Common Terminology Criteria for Adverse Events, Version 4.0. Participants were followed for 28 days after discontinuing treatment for safety and monitoring of AEs.
Time Frame: Median treatment duration in Phase 2 per group: Ewings Sarcoma = 14 weeks (3-31), Neuroblastoma = 7 weeks (3-23), Rhabdomyosarcoma = 5 weeks (1-13). Participants were followed for 28 days after discontinuing treatment for safety and monitoring of AEs.
Population: Safety Population: all participants who took at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Ewing's Sarcoma | Phase 2: Neuroblastoma | Phase 2: Rhabdomyosarcoma
Number analyzed (Participants) | 14 | 14 | 14
Participants
  TEAE | 14 | 14 | 14
  Treatment-related (TR) TEAE | 13 | 12 | 12
  Grade 3 or 4 TEAE | 12 | 13 | 12
  TR Grade 3 or 4 TEAE | 9 | 9 | 10
  Serious TEAE | 6 | 6 | 11
  TR Serious TEAE | 2 | 2 | 6
  TEAE Leading to Drug Discontinuation | 3 | 1 | 3
  TR TEAE Leading to Drug Discontinuation | 1 | 0 | 3
  TEAE Leading to Dose Reduction | 4 | 5 | 4
  TR TEAE Leading to Dose Reduction | 4 | 4 | 4
  TEAE Leading to Drug Interruption | 5 | 3 | 4
  TR TEAE Leading to Drug Interruption | 3 | 3 | 2
  TEAE Leading to Death | 0 | 2 | 3
  TR TEAE Leading to Death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Median treatment duration in Phase 1 was 7.0 weeks, with minimum and maximum duration of 1 and 49 weeks, respectively. Median treatment duration in Phase 2 per group: Ewings Sarcoma = 14 weeks (3-31), Neuroblastoma = 7 weeks (3-23), rhabdomyosarcoma = 5 weeks (1-13).
Description: All participants in both portions of the study were followed for 28 days after discontinuing treatment for safety and monitoring of AEs. AE's were analyzed in terms of TEAEs, which were defined as any AEs that began or worsened in severity on or after the start of study drug through 28 days after the last dose of study drug.
Groups:
- Phase 2: Nab-Paclitaxel 240 mg/m^2: Participants with Ewing's sarcoma, neuroblastoma, or rhabdomyosarcoma: nab-paclitaxel at the RP2D (240 mg/m^2 in participants weighing > 10 kg and 11.5 mg/kg in participants weighing ≤ 10 kg) IV on Days 1, 8 and 15 of a 28-day cycle until disease progression, death, withdrawal of consent, or unacceptable toxicity.
Arm/Group | Phase 1: Nab-Paclitaxel 120 mg/m^2 | Phase 1: Nab-Paclitaxel 150 mg/m^2 | Phase 1: Nab-Paclitaxel 180 mg/m^2 | Phase 1: Nab-Paclitaxel 210 mg/m^2 | Phase 1: Nab-Paclitaxel 240 mg/m^2 | Phase 1: Nab-Paclitaxel 270 mg/m^2 | Phase 2: Nab-Paclitaxel 240 mg/m^2
All-Cause Mortality (participants affected / at risk) | 14/16 | 7/8 | 11/14 | 5/11 | 8/8 | 5/7 | 25/42
Serious Adverse Events (participants affected / at risk) | 10/16 | 7/8 | 6/14 | 5/11 | 3/8 | 4/7 | 23/42
Other Adverse Events (participants affected / at risk) | 16/16 | 8/8 | 14/14 | 11/11 | 8/8 | 7/7 | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Nab-Paclitaxel 120 mg/m^2 (N=16) | Phase 1: Nab-Paclitaxel 150 mg/m^2 (N=8) | Phase 1: Nab-Paclitaxel 180 mg/m^2 (N=14) | Phase 1: Nab-Paclitaxel 210 mg/m^2 (N=11) | Phase 1: Nab-Paclitaxel 240 mg/m^2 (N=8) | Phase 1: Nab-Paclitaxel 270 mg/m^2 (N=7) | Phase 2: Nab-Paclitaxel 240 mg/m^2 (N=42)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 4
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 4
Generalised oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 2 | 3 | 1 | 2 | 6
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Slow speech (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Anuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Nab-Paclitaxel 120 mg/m^2 (N=16) | Phase 1: Nab-Paclitaxel 150 mg/m^2 (N=8) | Phase 1: Nab-Paclitaxel 180 mg/m^2 (N=14) | Phase 1: Nab-Paclitaxel 210 mg/m^2 (N=11) | Phase 1: Nab-Paclitaxel 240 mg/m^2 (N=8) | Phase 1: Nab-Paclitaxel 270 mg/m^2 (N=7) | Phase 2: Nab-Paclitaxel 240 mg/m^2 (N=42)
Anaemia (Blood and lymphatic system disorders) | 8 | 6 | 6 | 5 | 6 | 6 | 27
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 6 | 1 | 2 | 5 | 5 | 3 | 18
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 6 | 2 | 1 | 2 | 2 | 3 | 5
Neutropenia (Blood and lymphatic system disorders) | 7 | 4 | 6 | 8 | 7 | 6 | 23
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 1 | 2 | 4 | 8
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Ear swelling (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 3
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 5
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 3 | 2 | 3 | 2 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 4 | 3 | 3 | 6 | 2 | 1 | 10
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 4 | 3 | 4 | 2 | 8
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 2 | 0 | 2
Eructation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 6 | 3 | 2 | 4 | 2 | 3 | 10
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 2 | 8
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 8 | 3 | 2 | 3 | 3 | 1 | 14
Asthenia (General disorders) | 1 | 1 | 1 | 1 | 3 | 1 | 9
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 2
Fatigue (General disorders) | 3 | 3 | 4 | 4 | 2 | 0 | 2
General physical health deterioration (General disorders) | 0 | 1 | 1 | 1 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 3 | 2 | 1 | 1 | 0 | 8
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 6 | 3 | 5 | 5 | 4 | 2 | 14
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bacillus bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 1 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Recall phenomenon (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1 | 3 | 1 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 1 | 1 | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 4 | 0 | 1 | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 1
Candida test positive (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electroencephalogram abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Glucose urine present (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 0 | 1 | 2 | 2 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 5 | 1 | 1 | 1 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1 | 1 | 2 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 4 | 2 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 0 | 2 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2 | 0 | 3 | 1 | 17
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0 | 1 | 0 | 1 | 3
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 2
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 3 | 2 | 3 | 2 | 1 | 1 | 11
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 0 | 3 | 2 | 3
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Visual field defect (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 3 | 1 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 1
Enuresis (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 2
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Ketonuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Genital pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 4 | 3 | 0 | 6
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 2 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 4 | 5 | 3 | 2 | 6
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 2 | 2 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 7
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 1 | 1 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1 | 0 | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 7
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 1
Toxic erythema of chemotherapy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is more than one year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to ninety days. Investigator must delete confidential information before submission or defer publication to permit patent applications

DOCUMENTS (2):
  • Study Protocol (2016-07-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT01962103/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/03/NCT01962103/SAP_001.pdf